CLINICAL TRIAL: NCT06056453
Title: Interpersonal Psychotherapy in Adolescents With Polycystic Ovary Syndrome
Acronym: IPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Psychological Association (APA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20-3033
Record Dates: First submitted 2022-12-07; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Interpersonal Psychotherapy; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPT (Experimental): Participate in IPT 6-week intervention group.
  Interventions: Behavioral: Interpersonal Psychotherapy
- UC (No Intervention): Continue with usual care.

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — IPT group-virtual
  Arms: IPT

SUMMARY:
The main purpose of this study is to find out whether taking part in a group-based interpersonal psychotherapy (IPT) program designed to improve mood and lessen stress in girls with PCOS will improve depression, unhealthy eating behaviors, weight, and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PCOS duration > 3 months
* 12-17 years old
* BMI > 75th percentile
* CESD > 16

Exclusion Criteria:

* Weekly or bi-weekly therapy with licensed behavioral health provider
* Inability to speak, read, or write in English (teen)
* Major medical conditions
* HbA1c > 7.0%
* Hormonal contraception < 3 months
* Metformin < 3 months
* Antidepressants/psychotropic medications < 4 weeks

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies-Depression Scale | Baseline
  Depression symptoms will be assessed by the Center for Epidemiologic Studies-Depression Scale. Scores range from 1 to 4. The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Center for Epidemiologic Studies-Depression Scale | 6-Week Follow-Up Assessment
  Depression symptoms will be assessed by the Center for Epidemiologic Studies-Depression Scale. Scores range from 1 to 4. The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Center for Epidemiologic Studies-Depression Scale | 6-Month Follow-Up Assessment
  Depression symptoms will be assessed by the Center for Epidemiologic Studies-Depression Scale. Scores range from 1 to 4. The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.

SECONDARY OUTCOMES:
Emotional Eating Scale Adapted for Children | Baseline, 6-Week Follow-Up Assessment, 6-Month Follow-Up Assessment
  Disordered eating will be assessed by the Emotional Eating Scale Adapted for Children. The scale has been adapted for children and assesses eating in response to negative affect, such as feeling sad or irritated. The scale ranges from "I have no desire to eat" to "I have a very strong desire to eat" and averages how many days a week the participant eats based on that feeling.
Loss-of-Control Eating Disorder Questionnaire | Baseline, 6-Week Follow-Up Assessment, 6-Month Follow-Up Assessment
  Loss-of-control eating will be assessed via the 19-item Loss-of-Control Eating Disorder Questionnaire (LOC-ED-Q), which shows sound psychometric properties in adolescents using Yes/No.
Reward Based Eating Drive Scale | Baseline, 6-Week Follow-Up Assessment, 6-Month Follow-Up Assessment
  Reward based eating will be assessed by the Reward Based Eating Drive Scale. This is a self-report questionnaire which assesses reward-based eating that shows sound psychometric properties. The total score is summed at the end; a higher total is indicative of reward-based eating.
BMI | Baseline, 6-Week Follow-Up Assessment, 6-Month Follow-Up Assessment
  Fasting BMI (kg/m2) will be derived from measured height in triplicate by stadiometer and measured fasting weight by calibrated digital scale. BMI z-score and BMI %ile will be computed to determine eligibility (BMI ≥75th percentile).
Insulin Resistance | Baseline, 6-Week Follow-Up Assessment, 6-Month Follow-Up Assessment
  Blood will be sampled via a venipuncture procedure following a 10-hour overnight fast to measure fasting insulin. Insulin resistance will be estimated from fasting insulin and glucose with the homeostatic model assessment of insulin resistance (HOMA-IR).
Dysglycemia | Baseline, 6-Week Follow-Up Assessment, 6-Month Follow-Up Assessment
  Blood will be sampled via a venipuncture procedure following a 10-hour overnight fast to measure fasting insulin. Insulin resistance will be estimated from fasting insulin and glucose with the homeostatic model assessment of insulin resistance (HOMA-IR).
Dyslipidemia | Baseline, 6-Week Follow-Up Assessment, 6-Month Follow-Up Assessment
  Blood will be sampled via a venipuncture procedure following a 10-hour overnight fast to measure dyslipidemia. Insulin resistance will be estimated from fasting insulin and glucose with the homeostatic model assessment of insulin resistance (HOMA-IR).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Gulley, PhD, Principal Investigator — Colorado State University
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided